CLINICAL TRIAL: NCT03460652
Title: A Multicenter, Dose-Optimized, Open-Label Safety Study With KP415 in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: KP415 Open-Label Safety Study in Children (6-12 Years of Age) With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zevra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP415.S01
Record Dates: First submitted 2018-02-12; First posted 2018-03-09 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2020-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — serdexmethylphenidate and dexmethylphenidate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label KP415 (Experimental): KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
  Interventions: Drug: KP415 oral capsule

INTERVENTIONS:
Drug: KP415 oral capsule — Once-daily oral dose
  Other Names: Azstarys; SDX/d-MPH

SUMMARY:
This study is a multicenter, dose-optimized, open-label safety study with KP415 in children with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
The study will consist of a Screening Period, a Dose Optimization Phase, and a Treatment Phase and a Follow-Up Visit, as follows:

* Screening Period: Subjects will undergo a screening period up to 30 days prior to entering the Dose Optimization Phase.
* Dose Optimization Phase: During the Dose Optimization Phase, subjects will be titrated to doses of 20, 30 or 40 mg KP415 based on tolerability and best individual dose-response in the opinion of the Investigator.
* Treatment Phase: Eligible subjects will receive single daily doses of KP415 for up to approximately 360 days (up to approximately 12 months). The dose of KP415 given in the Treatment Phase will be the dose of KP415 at the end of the Dose Optimization Phase. During the Treatment Phase, the dose of KP415 may be changed based on individual tolerability and best dose response (to either 20, 30, or 40 mg KP415 capsules). Safety, efficacy and sleep behavior assessments will be performed.
* Follow-Up Visit: 3 ±2 days after administration of the last dose of the Treatment Phase, subjects will enter a Follow-Up Visit to evaluate safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactive/impulsive presentation) per clinical evaluation and confirmed by the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
2. Subject must have a score of at least 3 (mildly ill) on the clinician-administered Clinical Global Impressions-Severity (CGI-S) scale.
3. Subjects who completed the efficacy study with KP415 may be rolled over into the current study.
4. Subject, subject's parent/legal guardian and caregiver (if applicable) must understand and be willing and able to comply with all study procedures and visit schedule.

Exclusion Criteria:

1. Subject with any clinically significant chronic medical condition that may interfere with the participant's ability to participate in the study.
2. Subject has any diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, any history of psychosis, autism spectrum disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances.
3. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood, or history of persistent neurological symptoms attributable to serious head injury.
4. Subject has a current (last month) psychiatric diagnosis other than specific phobia, motor skills disorders, oppositional defiant disorder, sleep disorders, elimination disorders, adjustment disorders, learning disorders, or communication disorders. Participants with school phobia or separation anxiety will not be eligible.
5. Subject has clinically significant suicidal ideation/behavior, based on a history of attempted suicide and the C-SSRS assessment at Screening or at any time before the last dose of study drug.
6. Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism, or excretion of study drug.
7. Subject has a history or presence of abnormal ECGs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (19):
- United States (19):
  - Woodland International Research, Little Rock, Arkansas
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Meridien Research, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Meridien Research, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Houston Clinical Trials, Houston, Texas

REFERENCES:
- [Derived] Childress AC, Cutler AJ, Patel M, Oh C. Analysis of Growth Velocity in Children with Attention-Deficit/Hyperactivity Disorder Treated for up to 12 Months with Serdexmethylphenidate/Dexmethylphenidate. J Child Adolesc Psychopharmacol. 2023 May;33(4):134-142. doi: 10.1089/cap.2023.0012. PMID 37204277
- [Derived] Childress AC, Marraffino A, Cutler AJ, Oh C, Brams MN. Safety and Tolerability of Serdexmethylphenidate/Dexmethylphenidate Capsules in Children with Attention-Deficit/Hyperactivity Disorder: A 12-Month, Open-Label Safety Study. J Child Adolesc Psychopharmacol. 2023 Mar;33(2):51-58. doi: 10.1089/cap.2022.0076. Epub 2023 Feb 20. PMID 36809150

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment: Optimized dose of KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
Period: Overall Study
Arm/Group | Active Treatment
Started | 282
Entered Treatment Phase (Treatment Phase Safety Population, which includes all enrolled subjects who received at least 1 dose of study medication and had at least 1 post-dose safety assessment in the Treatment Phase) | 238
Completed | 155
Not Completed | 127

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45
  Not Hispanic or Latino | 193
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 111
  White | 113
  More than one race | 9
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs will be assessed starting following the first dose of study drug, and ending with the Follow-Up Visit or Early Termination Visit.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment-Phase Safety Population: Optimized dose of KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
Arm/Group | Treatment-Phase Safety Population
Number analyzed (Participants) | 238
Participants
  Subjects with at least 1 TEAE | 143
  Subjects with a related TEAE | 108
  Subjects with a TEAE leading to discontinuation of study drug | 6
  Subjects with an SAE | 2
  Subjects with an AE leading to death | 0

2. Secondary Outcome: Change From Baseline in ADHD-RS-5 Total Score
Description: The clinician-administered ADHD-RS-5 is an 18-item scale that rates ADHD symptoms on a 4-point scale. Each item is scored using a combination of severity and frequency ratings from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe symptoms or a frequency of very often), so that the total ADHD-RS-5 scores range from 0 to 54. The 18 items can be divided into two 9-item subscales: One for hyperactivity/impulsivity and the other for inattentiveness.
Time Frame: Up to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Open-Label KP415: Optimized dose of KP415 (serdexmethylphenidate [SDX] Cl/ d-methylphenidate [d-MPH] HCl) oral capsule:
  28/6 mg SDX/d-MPH (molar equivalent to 20 mg d-MPH HCl), 42/9 mg SDX/d-MPH (molar equivalent to 30 mg d-MPH HCl), 56/12 mg SDX/d-MPH (molar equivalent to 40 mg d-MPH HCl)
Arm/Group | Open-Label KP415
Number analyzed (Participants) | 225
score on a scale | -29.0 (11.21)

3. Secondary Outcome: Change From Baseline in CGI-S
Description: The CGI-S is a clinician-rated scale that evaluates the severity of psychopathology (ADHD symptoms in this study) on a scale from 1 (not at all ill) to 7 (among the most severely ill).
Time Frame: Up to 12 months
Population: The Overall Efficacy Population was comprised of 225 subjects. Due to early terminations, 223 subjects remained at Visit 6 (Day 30) and 153 subjects remained at Visit 17 (Day 360)
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label KP415
Number analyzed (Participants) | 225
Participants
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 1 = Normal, not at all | 0
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 2 = Borderline mentally ill | 0
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 3 = Mildly ill | 5
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 4 = Moderately ill | 82
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 5 = Markedly ill | 112
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 6 = Severely ill | 26
  Baseline (Visit 2 for new subjects and Visit 5 for roll-over subjects): 7 = Among the most extremely ill patients | 0
  Visit 17 (Day 360): number analyzed (Participants) | 153
  Visit 17 (Day 360): 1 = Normal, not at all | 47
  Visit 17 (Day 360): 2 = Borderline mentally ill | 45
  Visit 17 (Day 360): 3 = Mildly ill | 52
  Visit 17 (Day 360): 4 = Moderately ill | 7
  Visit 17 (Day 360): 5 = Markedly ill | 1
  Visit 17 (Day 360): 6 = Severely ill | 1
  Visit 17 (Day 360): 7 = Among the most extremely ill patients | 0

4. Secondary Outcome: Change From Baseline in Children's Sleep Habits Questionnaire
Description: The modified, abbreviated Children's Sleep Habits Questionnaire (CSHQ) will be used to assess the sleep behavior. The CSHQ is a retrospective, 33-item parent questionnaire to examine sleep behavior in small children. Items are rated on a 3-point scale of "Usually", "Sometimes" and "Rarely" for occurrences in a number of key sleep domains: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness. Scores range from 33-99, with higher scores represent more disturbed sleep. Scores were obtained during a clinician-directed interview with the parent/guardian/caregiver.
Time Frame: Up to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-Label KP415
Number analyzed (Participants) | 228
score on a scale | -4.3 (5.20)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/238
Serious Adverse Events (participants affected / at risk) | 3/238
Other Adverse Events (participants affected / at risk) | 143/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=238)
exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (7) — asthma, status asthmaticus, bronchospasm, acute respiratory failure, hyperglycaemia
seizure (Nervous system disorders) | 1 (1)
aggression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=238)
psychiatric disorders (Psychiatric disorders) | 55
infections and infestations (Infections and infestations) | 67
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 46
investigations (Investigations) | 33
gastrointestinal disorders (Gastrointestinal disorders) | 19
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 15
nervous system (Nervous system disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03460652/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03460652/SAP_002.pdf